CLINICAL TRIAL: NCT06320652
Title: Implementation and Evaluation of Telemedicine in Cardiac Rehabilitation - a Study on Health Literacy, Health Related Quality of Life, and Family Support
Brief Title: Implementation and Evaluation of Telemedicine in Cardiac Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Nina Cecilie Tjustrup, PhD student, MSc, RN, Copenhagen University Hospital, Hvidovre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CUHospital
Record Dates: First submitted 2024-03-11; First posted 2024-03-20 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Rehabilitation
Keywords: Cardiac rehabilitation; Telemedicine; Video consultation; Home monitoring

STUDY DESIGN:
Intervention Model Description: First, all willing patients who are offered cardiac rehabilitation will comprise the control group. Following a period of implementing the adapted co-created cardiac telerehabilitation intervention. Patients in the control group have access to standard care at the cardiac outpatient clinic program comprising standard center-based cardiac rehabilitation. Patients in the intervention group will, in addition to standard care, be offered an individually tailored family-focused cardiac telerehabilitation developed through a co-creative process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (No Intervention): All willing patients who are offered cardiac rehabilitation will comprise the control group. Patients in the control group will have access to standard care at the cardiac outpatient clinic program comprising standard center-based cardiac rehabilitation. The cardiac outpatient clinic registers activities and monitors patient participation in cardiac rehabilitation. Data on patient demographic, diagnoses, educational backgrounds, civil status, and patient-reported outcomes will be collected from self-reported questionnaires at baseline, and 3 months after.
  The family members attendig the patients cardiac rehabilitation will recive a questionnaire on support fra the outpatient clinic nurses 3 months after the first consultation.
- Cardiac Telerehabilitation (Experimental): Patients in the intervention group will, in addition to standard care, be offered an individually tailored family-focused cardiac telerehabilitation (video consultations and home monitoring) developed through a co-creative process.
  The cardiac outpatient clinic registers activities and monitors patient participation in cardiac rehabilitation. Data on patient demographic, diagnoses, educational backgrounds, civil status, and patient-reported outcomes will be collected from self-reported questionnaires at baseline, and 3 months after the intervention.
  The family members attendig the patients cardiac rehabilitation will recive a questionnaire on support fra the outpatient clinic nurses 3 months after the first consultation.
  Interventions: Other: Cardiac telerehabilitation (video consultation and home monitoring)

INTERVENTIONS:
Other: Cardiac telerehabilitation (video consultation and home monitoring) — Patients with cardiac disease and earlier experiences with cardiac rehabilitation, family members, and nurses in the Departments of Cardiology at Amager and Hvidovre Hospital will be invited to work in a partnership and through a course of innovative co-creative workshops. It is recommended that usability studies have 5-15 participants, which is why we plan to enroll 3 cardiac patients, 3 relatives and 3 nurses from the outpatient clinic. Through the workshops, a rehabilitation program offering cardiac telerehabilitation will be co-created to comply with the preferences and perspectives of patients and family members and nurses from the outpatient clinic. Through these workshops we will learn which important components and elements should be prioritized when offering cardiac telerehabilitation (how, when, and why?).
  Arms: Cardiac Telerehabilitation

SUMMARY:
The overall aim is to develop and test the effect of a tailored patient and family focused cardiac tele rehabilitation intervention on health literacy by comparing it to standard care. Furthermore, to evaluate health-related quality of life, family support, and how the patients experience the communication and relationship with outpatient clinic nurses.

DETAILED DESCRIPTION:
The project is designed inspired by The Complex Intervention Framework (MRC-Guidelines) combined with a patient and family participatory design. The project will consist of three sub-studies. The first study is a co-creation development of a model for the cardiac telerehabilitation intervention. The second study is a quasi-experimental study with a quantitative comparison of the group receiving the cardiac telerehabilitation intervention and control group. The third study will be a descriptive qualitative study which aim to investigate patient's experience with CTR using participant observation and individual interview or dyadic interview.

ELIGIBILITY:
Inclusion Criteria:

* Patients and their family members affiliated with the Department of Cardiology at Amager and Hvidovre Hospital and attending cardiac rehabilitation.
* Patients diagnosed with ischemic heart disease, heart failure, persistent atrial fibrillation, and cardiac valve surgery.

Exclusion Criteria:

* Patients with substantial language barriers and limited cognitive function.
* Patients who can't use a smart phone, tablet, or computer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Health Literacy Questonnaire | 3 months
  Health literacy is investigated through instruments such as the Health Literacy Questionnaire (HQL).
  The HLQ contains 44 qustions that cover nine conceptually distinct areas of Health Literacy. Response options for each scale are determined by the content and nature of the items. For scale 1-5 four point ordinal response options are used (strongly disagree, disagree, agree and strongly agree), while for scales 6-9 five-point ordinal response options are used (cannot do, very difficult, quite difficult, quite easy and very easy).
  HLQ scale scores are calculated as unit-weighted sums of the constituents items averaged by the number of items in the scale such that the nominal range of the scale scores are 1-4 for scale 1-5 and 1-5 for scale 6-9. A low score means worse outcome and a high score means better outcome.

SECONDARY OUTCOMES:
The European Quality of life five dimensions questionnaire | 3 months
  The European Quality of life (EQ-5D-5L) questionnaire is a well-known generic and validated instrument for measuring health related quality of life, and it is used in a population health surveys, clinical trials and health economics evaluations.
  The EQ-5D-5L have five response levels in each dimensions (none, slight, modrate, severe and extreme problems). The EQ-5D-5L health ranges from 11111 corresponding full health to 55555 corresponding the worse health state. The The EQ-5D also include a EQ VAS 0-100 where the 0 is labelled the worst health state and 100 is labelled the best health state.
The Iceland-Family Perceived Support Questionnaire | 3 months
  The Iceland-Family Perceived Support Questionnaire (ICE-FPSQ) measures patients and families perceived support from nurses during and after meeting the health care system.
  The ICE-FPSQ has 14 qustions and scores range from minimum score of 14 points to a maximum of 70 points on two areas of perceived family support (Cognitive support (5 items) and Emotional support (9 items). Qustions are answered on a five-point Likert scale ranging from 1 (almost never) to 5 (all the time). A high score closer to 70 indicates a positive score.
The eHealth Literacy Questionnaire | 3 months
  The eHealth Literacy Questionnaire (eHLQ) consist of seven domains. Each item is scored using af four point ordinal scale, response options: strongly disagree, disagree, agree and strongly agree.
  eHLQ scale scores are calculated as unit-weighted sums of the constituents items averaged by the number of items in the scale such that the nominal range of the scale scores are 1-4. A low score means worse outcome and a high score means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Stine M Rosenstroem, Post.doc, Principal Investigator — Amager Hvidovre Hospital
Locations (1):
- University Hospital Amager and Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tjustrup NC, Rosenstrom S, Risom SS, Hove JD, Brodsgaard A. Developing a Cardiac TeleRehabilitation model using co-production with patients, family members, and healthcare professionals. Eur J Cardiovasc Nurs. 2026 Jan 21:zvag020. doi: 10.1093/eurjcn/zvag020. Online ahead of print. PMID 41559760
- [Derived] Rosenstrom S, Cecilie Tjustrup N, Kallemose T, Risom SS, Hove JD, Brodsgaard A. Evaluating a co-created model for video consultations in cardiac rehabilitation: impact on health literacy, quality of life and family support-a study protocol. BMJ Open. 2025 Oct 2;15(10):e101099. doi: 10.1136/bmjopen-2025-101099. PMID 41043840